CLINICAL TRIAL: NCT06404372
Title: A Pivotal, Blinded Multi-Center Study to Show the Safety and Effectiveness of the Demetech Barbed PDO Suture
Brief Title: To Show the Safety and Effectiveness of the Demetech Barbed Polydioxanone (PDO) Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sutura Medical Technology LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF-CLT-PRT
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Wrinkle
Keywords: Suture; Sutura; Demetech Barbed PDO Suture; Novathreads

STUDY DESIGN:
Masking Description: There will be a panel of the three evaluators who will be blinded. The treating physician, study staff, and office staff do not inform the panel of three blinded evaluators of whom they are viewing or of the chronological timepoint of the photograph.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Demetech Barbed PDO Suture (Experimental): Subjects who meet Inclusion/Exclusion criteria will receive treatment with Demetech Barbed PDO Sutures. Fifty-seven subjects will be treated. In addition, up to 2 run-in subjects may be treated with Demetech Barbed PDO Sutures by the investigator to allow the investigator to become familiar with Demetech Barbed PDO Suture characteristics. This run-in cohort will be required to meet all study inclusion/exclusion criteria and will be followed in the same manner as the non-run-in cohort.
  Interventions: Device: Demetech Barbed PDO Suture

INTERVENTIONS:
Device: Demetech Barbed PDO Suture — The Demetech Barbed PDO Suture will be used for the correction of midface wrinkles in all patients enrolled in this study.

SUMMARY:
The clinical trial, sponsored by Sutura Medical Technology, Inc., is a pivotal, blinded, multi-center study assessing the safety and effectiveness of the Demetech Barbed PDO Suture, an absorbable Polydioxanone suture, for the temporary treatment of midface wrinkles. The trial will enroll 57 subjects across up to four sites, following them over a 12-month period to evaluate improvements in wrinkles based on the Lemperle Classification Facial Wrinkle Scale. Primary endpoints include assessing the rate of adverse events and a significant reduction in wrinkle severity at 6 months, with secondary endpoints focusing on longer-term results and patient satisfaction.

DETAILED DESCRIPTION:
The study will be a pivotal, blinded, multi-center study to evaluate the safety and effectiveness of Demetech Barbed PDO Suture for the treatment of mid face wrinkles. Subjects who meet Inclusion/Exclusion criteria will receive treatment with Demetech Barbed PDO Sutures. Fifty-seven subjects will be treated. In addition, up to 2 run-in subjects may be treated with Demetech Barbed PDO Sutures by the investigator to allow the investigator to become familiar with Demetech Barbed PDO Suture characteristics. This run-in cohort will be required to meet all study inclusion/exclusion criteria and will be followed in the same manner as the non-run-in cohort.

Primary effectiveness will be assessed at 6 months. All subjects will be followed for a minimum of 12 months after treatment. Subjects will be followed up for safety via telephone or email at 72 hours after receiving treatment.

The primary effectiveness endpoint will be determined by the proportion of subjects with ≥1 point improvement on the Lemperle Classification of Facial Wrinkles Scale at 6 months compared to baseline as rated by a panel of three blinded evaluators. The Lemperle Scale will be used for photographic assessment by the blinded panel. Assessment of the secondary effectiveness endpoints will include the use of the Lemperle Scale by photograph by the blinded panel and live by the Investigator, as well as Investigator- and Subject-rated GAIS, and FACE-Q.

Safety will be assessed at each follow-up visit. Subjects will be seen for follow up visits at 2 weeks, 6 weeks, 3 months, 6 months, 9 months, and 12 months from treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 22+ years of age.
2. Subject received a rating, in each cheek, by PI of at least Class 1 or more for wrinkling in the midface according to the Lemperle Scale Classification of Facial Wrinkling.
3. If a woman is of childbearing potential (not amenorrheic for the previous 24 months or not surgically sterile), then she must have a confirmed negative urine pregnancy test result at screening. If treatment is not provided at the screening visit, a negative urine pregnancy test result is required within 7 days before treatment.
4. If a woman of childbearing potential, subject confirms she will utilize at least one form of contraception throughout the duration of the study.
5. Subjects who desire cheek lifting to correct age-related wrinkles in the midface as recommended by the treating investigator.
6. Subjects who are able to understand the study requirements, including the obligation not to receive any other facial procedures or treatments affecting mid-face at any time during the study.
7. Subjects who are willing to participate in the study and to sign a witnessed/informed consent form.
8. Subjects who are logistically able to present for all study visits and meet all study requirements.
9. Subjects who are willing to complete the 30-day diary.
10. Subjects who pass the pinprick and/or cotton swab facial nerve assessment.

Exclusion Criteria:

1. Abnormal rating in midface sensation, with inability to feel a 0.4 G monofilament or a cotton wisp at any site on the midface.
2. Active acne or prominent acne scars in the treatment area.
3. Active inflammatory or infectious conditions.
4. Allergy or foreign body sensitivities to plastic biomaterials.
5. Known bleeding disorder.
6. Breastfeeding, pregnant, or not on/willing to use contraception if of childbearing potential.
7. Collagen skin disorder.
8. Pre-existing facial asymmetry.
9. History of any device use on the mid-face in the prior 6 months (e.g., laser, IPL, radiofrequency, ultrasound, micro-needling, micro needle radiofrequency, or cool based treatments).
10. History of autoimmune or connective tissue disease.
11. History of facelift, midface lift, lower facelift, or neck lift that changes the facial structure and anchor points.
12. History of fat transfer to the midface.
13. History of injectable fillers other than temporary fillers such as Hyaluronic Acid (HA) or Radiesse to the midface at any time. Permanent and semi-permanent fillers are not allowed (e.g., Poly-L-lactic acid (PLLA), Sculptra).
14. History of Kybella in the prior 6 months.
15. History of facial trauma in the mid-face.
16. History of facial surgical procedures.
17. Inability to chew, puff cheek, or smile broadly.
18. Metabolism irregularities.
19. On immunosuppressive therapy.
20. Recent weight loss or intention to lose a significant amount of weight during the study period (2 BMI Points).
21. Subjects who have undergone cosmetic facial plastic surgery (with the exception of rhinoplasty or upper blepharoplasty, more than 2 years prior to enrollment), tissue grafting, or tissue lifting or augmentation with any permanent or semi-permanent filler.
22. Subjects who have had temporary facial dermal filler injections below the orbital rim with HA-based fillers or Radiesse within 18 months, porcine-based collagen fillers within 24 months, or neuromodulator injections to the midface or lateral canthal lines, mesotherapy, or resurfacing (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, chemical peel, or other ablative or non-ablative procedures) within 6 months of entry in the study or who were planning to undergo any of these procedures at any time during the study.
23. Subjects who have very thin skin in the mid-face region, who have the tendency to accumulate fluid in the lower eyelids, or who have large infraorbital fat pads.
24. Subjects who have mid-face volume deficit due to congenital defect, trauma, abnormalities in adipose tissue related to immune-mediated diseases such as generalized lipodystrophy, partial lipodystrophy (e.g., Barraquer-Simons syndrome), inherited disease, or HIV-related disease.
25. Subjects who have serious concurrent illness which may lead to problems with wound healing (e.g., uncontrolled diabetes or vascular disease).
26. Subjects with known or suspected family history of problems with keloid scarring.
27. Subjects with serious neurological or psychological conditions which could prevent the subject from cooperating with treatment or post-procedure care and assessment.
28. Smokers, since this may compromise wound healing.
29. Subjects who have a current or prior history within the last 3 years of neoplasm and/or any active neoplasm in the face or that in the opinion of the Investigator may make them not a suitable candidate.
30. Subjects currently enrolled in other clinical trials.
31. Subjects taking Warfarin or other anticoagulants. These subjects may experience a significant risk of problems with post-operative bleeding.
32. Subjects who have taken, in the last 2 weeks, ad-lib medication or herbal supplements that may increase risk of bleeding. This includes aspirin or other herbal supplements known to increase risk of bleeding.
33. Subjects with significant co-morbidities (e.g., heart disease, strokes, or angina) that in the opinion of the Investigator may prevent the subject from completing the study.
34. Subjects with planned cosmetic procedures, facial or dental surgery during the follow-up period.
35. Other concerning health issue in the opinion of the Investigator.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Improvement from Baseline on the Lemperle Classification Wrinkle Scale | 6 Month
  The primary effectiveness endpoint is the proportion of subjects with ≥1 point improvement on the Lemperle Classification Facial Wrinkle Scale at 6 months compared to baseline, as rated by a panel of three blinded evaluators. The median score as rated by the blinded panel using subject photographs will be used to determine if a subject is a responder. Clinical effectiveness will be demonstrated by superiority of this 6-month response rate over a target rate of 60%

SECONDARY OUTCOMES:
Proportion of Subjects with ≥1 Point Change from Baseline on the Lemperle Classification Facial Wrinkle Scale | 3, 9, and 12 Months
  Individual endpoints at each timepoint of 3, 9, and 12 months for the proportion of subjects with ≥1 point change from baseline on the Lemperle Scale, as rated by a panel of three blinded evaluators. The Lemperle Scale is a 6-point wrinkle classification scale with classification values of 0 to 5 wherein the higher value indicates more severe wrinkles, which are considered worse outcomes.
Change from Baseline on the Lemperle Classification Facial Wrinkle Scale as rated by a panel of three blinded evaluators | 3, 6, 9, and 12 Months
  Change from baseline at each timepoint of 3, 6, 9, and 12 months on the Lemperle Scale, as rated by a panel of three blinded evaluators. The Lemperle Scale is a 6-point wrinkle classification scale with classification values of 0 to 5 wherein the higher value indicates more severe wrinkles, which are considered worse outcomes.
Proportion of Subjects with ≥1 Point Change from Baseline on the Lemperle Classification Facial Wrinkle Scale | 3, 6, 9, and 12 Months
  Individual endpoints at each timepoint of 3, 6, 9, and 12 months for the proportion of subjects with ≥1 point change from baseline on the Lemperle Scale, as rated by the Investigator. The Lemperle Scale is a 6-point wrinkle classification scale with classification values of 0 to 5 wherein the higher value indicates more severe wrinkles, which are considered worse outcomes.
Change from Baseline on the Lemperle Classification Facial Wrinkle Scale as rated by the Investigator | 3, 6, 9, and 12 Months
  Change from baseline at each timepoint of 3, 6, 9, and 12 months on the Lemperle Scale, as rated by the Investigator. The Lemperle Scale is a 6-point wrinkle classification scale with classification values of 0 to 5 wherein the higher value indicates more severe wrinkles, which are considered worse outcomes.
Change in Investigator-rated Global Aesthetic Improvement Scale (GAIS) | 6 Weeks, 3, 6, 9, 12 Months
  Individual endpoints at each timepoint of 6 weeks, 3, 6, 9, and 12 months for change in Investigator-rated. The GAIS) is a 7-point scale with values of -3 to 3 wherein the higher value indicates a greater degree of change in aesthetic appearance.
Change in Subject-rated Global Aesthetic Improvement Scale | 6 Weeks, 3, 6, 9, 12 Months
  Individual endpoints at each timepoint of 6 weeks, 3, 6, 9, and 12 months for change in Subject-rated GAIS. The GAIS) is a 7-point scale with values of -3 to 3 wherein the higher value indicates a greater degree of change in aesthetic appearance.
FACE-Q Appraisal of Cheeks and Age Appraisal Questionnaires Satisfaction with Cheeks and Age Appraisal scales as rated by the Subject. | 6 Weeks, 3, 6, 9, 12 Months
  Individual endpoints at each timepoint of 6 weeks, 3, 6, 9, and 12 months for change from baseline on each of the validated FACE-Q Satisfaction with Cheeks and Age Appraisal scales as rated by the Subject.

CONTACTS AND LOCATIONS:
Overall Officials: Sherly Soleiman, MD, Principal Investigator — Cosmetic Injectables Center; Chaitali Nangrani, MD, Principal Investigator — Vedas Med Spa; Kristin Tarbet, MD, Principal Investigator — Dr. Kristin Tarbet Facial Plastic Surgery; Amit Kocher, MD, Principal Investigator — Rejuva Medical Aesthetics
Locations (4):
- United States (4):
  - Rejuva Medical Aesthetics, Los Angeles, California
  - Cosmetic Injectables Center, Sherman Oaks, California
  - Vedas Med Spa, The Woodlands, Texas
  - Dr. Kristin Tarbet Facial Plastic Surgery, Bellevue, Washington